CLINICAL TRIAL: NCT05441202
Title: The Efficacy of Transdermal Therapy for Lung nodule---an Real Word Observational Study
Brief Title: Lung Nodule Intervention Cohort Study
Acronym: LNICS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Chronic Respiratory Disease Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: LN002
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-01

CONDITIONS: Incident Lung Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: transdermal therapy — transdermal therapy with Chinese medicine

SUMMARY:
Incident lung nodule is quite common in China. The major treatment method is long-term floolow up without a specific intervention. We aim to investigate the efficacy an safty of a novel transdermal therapy with Chinese herb. The study included two arms: one arm is routine treatment and another arm is routine treatment plus transdermal therapy. The study end point is the change of lung nodule size under CT scan.

ELIGIBILITY:
Inclusion Criteria:

* incident lung nodule patients

Exclusion Criteria:

* severe baseline conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient with incident lung nodule after health check up
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
change of lung nodule size | three months minimal
  change of lung nodule size before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Guang An Men Hospital, Beijing, Beijing Municipality, China